CLINICAL TRIAL: NCT02786186
Title: A Registry of Patients With Moderate to Severe Chronic Plaque Psoriasis in Canada and Latin AmErica (LACan)
Brief Title: A Registry of Patients With Moderate to Severe Plaque Psoriasis
Acronym: PURE
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457ACA02
Record Dates: First submitted 2016-05-06; First posted 2016-05-30 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Chronic Plaque Psoriasis; Cosentyx; Secukinumab; Moderate to severe plaque psoriasis; PURE registry; Registry
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Secikinumab: Patients treated with secukinumab
  Interventions: Drug: Secikinumab
- Approved standard of care: Patients treated with other indicated therapies (systemic, phototherapy, or biologic therapy)
  Interventions: Drug: Secikinumab

INTERVENTIONS:
Drug: Secikinumab
  Other Names: AIN457

SUMMARY:
The main purpose of the current study will be to provide real - world evidence regarding the safety and effectiveness of secukinumab in the management of patients with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
PURE is a multi-national, prospective, observational cohort study of patients with moderate to severe chronic plaque psoriasis aimed at assessing the real-world safety and effectiveness of secukinumab and other indicated therapies. The study will enroll patients for whom, prior to and independent of study enrollment, the treating physician has decided to treat with secukinumab, or one of the other indicated therapies regimens approved for the management of moderate to severe chronic plaque psoriasis.

Two study cohorts will be defined by patients treated with secukinumab (Cohort 1), and patients treated with other indicated therapies (systemic, phototherapy, or biologic therapy; Cohort 2). Each investigator will recruit approximately the same number of patients in each treatment arm. 2,500 patients (1,250 patients in each cohort) will be followed over a period of 5 years from the Baseline assessment (Visit 1).

ELIGIBILITY:
Inclusion Criteria:

1. - Patients able to give written informed consent
2. - Patients at least 18 years of age at time of informed consent signature
3. - Confirmed diagnosis of chronic moderate to severe chronic plaque-type psoriasis diagnosed by a specialist and presence of moderate to severe psoriasis symptoms according to physician's clinical judgment at the time of recruitment.
4. - Patients initiating a treatment for psoriasis as per regional policy. This will include secukinumab, other biologics, systemic treatments, and phototherapy. Decision to treat with any of the above-mentioned treatments must have been reached prior to and independently of recruitment in the study.
5. - Treatments prescribed in accordance to the product monograph and regional regulatory and reimbursement policies
6. - Patients able to understand and communicate with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. - Unwillingness or inability to comply with the study requirements
2. - Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with moderate to severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 2384 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Change from Baseline through month 60
  Incidence of all adverse events in the study cohorts as measured by:
  1. The proportion of patients that experience at least one event;
     and
  2. The number of events per participant

SECONDARY OUTCOMES:
Percentage of Participants Achieving PASI 50/75/90/100 Response or IGA 0 or 1 Response | Change from Baseline through month 60
  PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section(head: 0.1, arms: 0.2 body: 0.3 legs: 0.4)
Mean change for Work Productivity and Activity Impairment (WPAI) score | Change from Baseline through month 60
Mean change for Hospital Anxiety and Depression Scale (HADS) score | Change from Baseline through month 60
Mean change for Psoriasis Symptom Diary (PSD) score | Change from Baseline through month 60
Mean change for Treatment Satisfaction Scale (TSS) score | Change from Baseline through month 60
Mean change for Dermatology Life Quality Index (DLQI) score | Change from Baseline through month 60
Mean change for Psoriasis Epidemiology Screening Tool (PEST) score | Change from Baseline through month 60
Mean change for direct and indirect cost associated to Psoriasis | Change from Baseline through month 60

CONTACTS AND LOCATIONS:
Locations (60):
- Argentina (6):
  - Novartis Investigative Site, Adrogué, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Canada (38):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Nanaimo, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Brandon, Manitoba
  - Novartis Investigative Site, Winnepeg, Manitoba
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Fredericton, New Brunswick
  - Novartis Investigative Site, Rothesay, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kentville, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Cobourg, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Nepean, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, North Bay, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Richmond Hill, Ontario
  - Novartis Investigative Site, Stoney Creek, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
  - Novartis Investigative Site, Sainte Hyacinthe, Quebec
  - Novartis Investigative Site, Verdun, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, San José, Costa Rica
- Dominican Republic (2):
  - Novartis Investigative Site, Santiago de los Caballeros
  - Novartis Investigative Site, Santo Domingo
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, Ciudad de Guatemala
  - Novartis Investigative Site, Guatemala City
- Mexico (9):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Del Tlalpan, Mexico City
  - Novartis Investigative Site, Guadalajara Jalisco, Mexico
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Pedro Garza García, Nuevo León
  - Novartis Investigative Site, Toluca, State of Mexico
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Mexico City
- Novartis Investigative Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Papp KA, Gooderham M, Dei-Cas I, LopezTello A, Garcia-Rodriguez JC, Taveras CY, Rousselin AH, Lavieri A, Maiolino M, Quintero DGV, Rihakova L, Salibe M, Pertuz W. Effectiveness and Safety of Secukinumab in Latin American Patients with Moderate to Severe Plaque Psoriasis: PURE Registry 12-Month Data. Dermatol Ther (Heidelb). 2023 Jan;13(1):269-283. doi: 10.1007/s13555-022-00849-0. Epub 2022 Dec 10. PMID 36496547
- [Derived] Papp KA, Gooderham M, Beecker J, Lynde CW, Delorme I, Dei-Cas I, Albrecht L, Rampakakis E, Sampalis JS, Vieira A, Hussein S, Chambenoit O, Rihakova L. Rationale, objectives and design of PURE, a prospective registry of patients with moderate to severe chronic plaque psoriasis in Canada and Latin America. BMC Dermatol. 2019 Jun 21;19(1):9. doi: 10.1186/s12895-019-0087-3. PMID 31226985